CLINICAL TRIAL: NCT06758193
Title: Validity and Reliability of the The Measure of Activity Performance of the Hand Scale in Patients With Carpal Tunnel Syndrome
Brief Title: Validity and Reliability of the MAP-Hand Scale in Patients With Carpal Tunnel Syndrome
Status: Enrolling by invitation | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Atahan TURHAN, Lecturer Dr., Kirsehir Ahi Evran Universitesi
Other Study IDs: KAEU-T.ATAHAN-006
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: Carpal Tunnel Syndrome; Reliability; Validity
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group
  Interventions: Other: No intervention was applied in this study.

INTERVENTIONS:
Other: No intervention was applied in this study. — No intervention was applied in this study.

SUMMARY:
The primary aim of the study was to determine the validity and reliability of the "MAP-Hand (Measure of Activity Performance of the Hand)" scale in patients with carpal tunnel syndrome. The secondary aim of the study was to evaluate the hand activity performance in patients with carpal tunnel syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above and able to read and write
2. Diagnosed with mild or moderate unilateral CTS according to electroneuromyography results at least 6 months ago
3. Motor-sensory symptoms such as numbness and loss of strength in the hand for at least three months
4. Volunteers with no history of diabetes, no medical treatment or injections, no surgery, and no cervical radiculopathy or polyneuropathy

Exclusion Criteria:

1. Those with trauma, deformity, fracture, muscle contracture and atrophy in the shoulder, forearm and hand
2. Those who have received corticosteroid injections into the carpal tunnel area within the last three months and have been included in a physiotherapy program
3. Those who have cognitive problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who apply to the Physical Medicine and Rehabilitation Polyclinic with complaints of hand-wrist pain will be examined by a physical therapist. Patients who are diagnosed with Carpal Tunnel Syndrome through physical examination, meet the inclusion criteria, and agree to participate in the study will be included in the study.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Hand Activity Performance | 24 weeks
  The MAP-Hand (Measure of Activity Performance of the Hand) scale is a scale consisting of 18 items that evaluates the activity performance of the hand. These items are scored between 1 and 4 and the total score ranges from 18 to 72. Lower scores indicate better activity performance. The participants' hand activity performance will be evaluated with the MAP-Hand scale. The reliability and validity of the Turkish form of the MAP-Hand scale was conducted by Bayraktar and colleagues. However, their work has not yet been published. The necessary permissions have been obtained to use the scale.

SECONDARY OUTCOMES:
Grip Strength | 24 weeks
  Hand grip strength will be measured with a Camry brand digital dynamometer. Participants will be assessed in an upright position on a chair with their feet on the floor, with their arm next to their body, elbow in 90-degree flexion, forearm in midrotation and wrist in neutral. Participants were verbally encouraged during the test. Measurements were repeated three times and the highest value will be recorded in kilograms.
Pain | 24 weeks
  The participants' pain intensity during rest, activity and night will be measured with VAS. According to VAS, pain intensity is evaluated on a 10 cm line between 0 (no pain) and 10 (most severe pain). High scores indicate severe pain. Participants will be asked to indicate the intensity of pain they feel on a 10 cm scale.
Hand and Finger Skills | 24 weeks
  The participants' hand and finger skills will be tested with the 9-Hole Peg Test (9-DÇT). The 9-DÇT is a test that measures hand and finger skills in daily life. A pegboard with 9 holes, 3.2 cm wide, each hole 1.3 cm deep, will be placed in front of the participants in a way that it will be in the midline of the body. Participants will be asked to randomly place 9 wooden pins on the 9-hole pegboard as quickly as possible and then remove the pins from the pegboard one by one and put them in the box. At the end of 3 trials, the times will be recorded in seconds with a stopwatch and the shortest time will be recorded. A longer time to complete the test indicates inadequacy in hand-finger skills.
Hand Health Status | 24 weeks
  Hand health status will be assessed with the "Michigan Hand Outcome Questionnaire (MESA)". MESA consists of 37 questions and is a questionnaire with 6 parameters that evaluate general hand function, daily living activities, pain, work, aesthetics and satisfaction. Each question is evaluated with a 5-point Likert scale and a high score indicates a good status.
Carpal Tunnel Symptom Severity | 24 weeks
  The symptom severity and functional status of the participants will be evaluated with the "Boston Carpal Tunnel Syndrome Questionnaire (BCTQ)". BCTQ consists of the symptom severity scale (SSS) and the functional status scale (FSS) that evaluate the patient in two categories. While the SSS consists of 11 items, the FSS consists of 8 items. The average score is calculated by the ratio of the total score obtained to the number of questions. An increase in the average score indicates that the symptom is severe and functional limitation increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Kirsehir Ahi Evran University, Kırşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No